CLINICAL TRIAL: NCT04261413
Title: A Multicenter, Open Label, Two-step, Phase Ia/Ib Study of Tumor Targeted Prodrug RS-0139 in Patients with a Recurrent, Locally Advanced or Metastatic Solid Tumors
Brief Title: Phase Ia/Ib Study of RS-0139 in Patients with a Recurrent, Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RS Arastirma Egitim Danismanlik Ilac Sanayi Ticaret A.S. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS-001
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumors
Keywords: solid tumors; chemotherapy; targeted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RS-0139 (Experimental): There will be only RS-0139 arm in the study.
  Interventions: Drug: RS-0139

INTERVENTIONS:
Drug: RS-0139 — RS-0139 will be administered for the indication of solid tumors.

SUMMARY:
This study designed as a multicenter, open label, two-step study to determine the optimum dose, pharmacokinetics, and the safety of RS-0139 in patients with a recurrent, locally advanced or metastatic solid tumors. The research is planned as a two-step study (Phase Ia and phase Ib) and accelerated titration design (ATD) is used.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have consented to participation in the trial.
* Patients of both sexes aged between 18 and 75 years.
* Patients with relapsed or refractory solid tumors who have failed available standard therapy or are not candidates for standard therapy.
* Patients who are willing to provide fresh or archival biopsy material before their participation to identify the integrin expression levels (for Phase Ib only).
* Patients who completed the previous treatments 21 days before the first dose of the study drug.
* Patients who have at least three months of life expectancy.
* Patients with ECOG performance score 0 to 1.
* Patients with adequate organ function defined as:

  * Hemoglobin ≥10 mg/dl
  * Neutrophil ≥1,500/µL
  * Platelet ≥100,000/µL
  * Creatinine ≤1.5xULN or creatinine clearance ≥60mL/sec/1.73m2
  * Total bilirubin ≤ 1.5xULN
  * AST/ALT ≤2.5xULN; for patients who have confirmed liver metastasis: AST/ALT ≤5xULN.
  * Prothrombin time ≤1.5xULN (in case of no anticoagulant treatment).
  * Normal levels of serum magnesium and potassium concentrations

Exclusion Criteria:

* Patients with active and/or uncontrolled central nervous system (CNS) metastasis.
* Patients who have interstitial lung disease or interstitial pneumonia.
* Patients who have serious cardiac dysfunction.
* Patients who have insufficient target organ function.
* Patients with positive tests for HAV, HBV, HCV or HIV.
* Patients who experienced grade 3 or higher toxicity related to the previous docetaxel treatment.
* Female patients who are pregnant or breastfeeding.
* Male patients with pregnant female partners.
* Patients enrolled in another clinical trial at the same time or recently completed an investigational drug study and received the last dose of an investigational drug within 30 days or five half-lives (whichever is longer).
* Patients who have serious medical conditions such as uncontrolled infection or untreated wounds.
* Patients who have bone marrow transplantation history.
* Patients who have hypersensitivity to docetaxel, components of RS-0139 and/or other taxanes.
* Patients taking inhibitors or inducers of CYP3A4, including grapefruit juice and OTC medications such as St. John's Wort.
* Patients who, in the judgment of the PI, are likely to be non-compliant or unable to cooperate.
* Patients who cannot be contacted in case of emergency.
* Patients who are the PI or sub-investigator, research assistant, pharmacist, study coordinator or other staff directly involved in conducting the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | At the end of each cycle (Each cycle is 21 days)
The incidence of AEs, serious adverse events (SAEs) and treatment-emergent adverse events (TEAEs). | At the end of each cycle (Each cycle is 21 days)

SECONDARY OUTCOMES:
Anti-tumor activity measured by tumor shrinkage (based on CT-scan evaluations) | At the end of Phase Ib (assessed up to 1 year)
Change in CA 125 / CA15-3 / CA 19-9 / CA 72-4 (depends on the tumor type) | At the end of Phase Ib (assessed up to 1 year)
Change in circulating tumor cells | At the end of Phase Ib (assessed up to 1 year)
Objective Response Rate (ORR) | At the end of Phase Ib (assessed up to 1 year)
Progression-Free Survival (PFS) | At the end of Phase Ib (assessed up to 1 year)
Duration of Response (DoR) | At the end of Phase Ib (assessed up to 1 year)
Peak plasma concentration (Cmax) | At the end of the Phase Ia and Ib (assessed up to 1 year)
AUC(o-t) | At the end of the Phase Ia and Ib (assessed up to 1 year)
AUC(0-∞) | At the end of the Phase Ia and Ib (assessed up to 1 year)
tmax | At the end of the Phase Ia and Ib (assessed up to 1 year)
t1/2 | At the end of the Phase Ia and Ib (assessed up to 1 year)
λz | At the end of the Phase Ia and Ib (assessed up to 1 year)
CL | At the end of the Phase Ia and Ib (assessed up to 1 year)
Vss | At the end of the Phase Ia and Ib (assessed up to 1 year)

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Abdurrahman Yurtaslan Ankara Onkoloji Eğitim ve Araştırma Hastanesi, Ankara
  - Koç University Hospital Phase I Center, Istanbul

IPD SHARING:
Plan to Share IPD: No